CLINICAL TRIAL: NCT03011931
Title: Simvastatin Metabolism as a Test for Celiac Disease Activity
Brief Title: Simvastatin Metabolism as a Test for CD Activity (IRB 15-007568]
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Entero Therapeutics (Industry)
Collaborators: Immunogenics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-007568
Record Dates: First submitted 2016-10-03; First posted 2017-01-06 (Estimated); Last update posted 2024-08-05 (Actual); Status verified 2020-01

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Simvastatin (Experimental): Simvastatin tablet, 20 mg, one time by mouth
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 20 mg Simvastatin given, Blood draw, Urine collection, Celiac serology testing, DNA sampling, Dietary review
  Other Names: Zocor

SUMMARY:
To study the correlation between simvastatin metabolism by the enterocyte and the histologic state of the intestine in treated celiac disease.

DETAILED DESCRIPTION:
A cross sectional design incorporating subjects with active celiac disease and healed celiac disease (based on clinically-obtained biopsies); and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Gluten-free diet for at least 1 year
2. Clinical endoscopy within the past month
3. Biopsies must show no villous atrophy or villous blunting
4. Villous height to crypt depth (VHCD) ratio measurement should be 2.5:1 or greater

Exclusion Criteria:

1. 1st degree relative with Celiac Disease
2. Positive tTG IgA, already on simvastatin or statin agent
3. Unable to stop non-steroidal or anti-inflammatory drugs
4. Prior history of GI surgery other than appendectomy or cholecystectomy
5. Taking drugs know to inhibit or activate CYP3A4
6. Unable to avoid food known to inhibit CYP3A4
7. History of a reaction to statin drugs in the past
8. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Compare simvastatin metabolism with intestinal biopsies | Within one month of visit

SECONDARY OUTCOMES:
Villous height and crypt depth | Within 1 month of visit
  As measured in intestinal biopsies
Dietary interview | At initial visit
  To determine whether the patient is strictly adherent, mostly adherent or non-adherent to a gluten-free diet
Urinalysis | Prior to administration of simvastatin and at the 3-hour mark
  Looking for traces of gluten peptides
Serologic testing | Prior to administration of simvastatin
  tTG IgA titer level determination
DNA sampling | Prior to administration of simvastatin
  Genetic testing associated with celiac disease (DQ2 and DQ8)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Murray, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Simvastatin Metabolism as a Test for Celiac Disease Activity - Mayo Clinic — https://www.mayo.edu/research/clinical-trials/cls-20304518